CLINICAL TRIAL: NCT04256473
Title: Dual Thrombolytic Therapy With Mutant Pro-urokinase (M-pro-urokinase, HisproUK) and Low Dose Alteplase for Ischemic Stroke
Brief Title: Dual Thrombolytic Therapy With Mutant Pro-urokinase and Low Dose Alteplase for Ischemic Stroke
Acronym: DUMAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: DUMAS is sponsored by an unrestricted grant from Thrombolytic Science International, paid to the institution. (Unknown)
Responsible Party: Principal Investigator, Nadinda van der Ende, PI: Prof. Dr. DWJ Dippel and A. van der Lugt, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DUMAS-1.1
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Ischemic Stroke
Keywords: Randomized Controlled Trial; Thrombolytic treatment; Intracranial hemorrhage; Mutant pro-urokinase; Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke; Intracranial Hemorrhages | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Bolus of IV alteplase (5 mg) followed by continuous infusion of HisproUK 40 mg/hr during 60 minutes.
  Depending on results of interim analyses, the alternate dose may be revised to a lower dose (30mg/hr during 60 minutes) or a higher dose (50mg/hr during 60 minutes).
  Interventions: Drug: mutant pro-urokinase
- Control (Active Comparator): Usual care with alteplase 0.9 mg/kg in 60 minutes
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: mutant pro-urokinase — Intravenous administration
  Other Names: HisproUK
  Arms: Intervention
Drug: Alteplase — Intravenous administration
  Other Names: Actilyse
  Arms: Control

SUMMARY:
Randomized controlled phase II trial to test the safety and preliminary efficacy of a dual thrombolytic treatment consisting of a small intravenous (IV) bolus of alteplase followed by IV infusion of mutant pro-urokinase against usual treatment with IV alteplase in patients presenting with ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of ischemic stroke;
* A score of at least 1 on the NIH Stroke Scale;
* CT ruling out intracranial hemorrhage;
* Treatment possible within 4.5 hours from symptom onset or last seen well;
* Meet the criteria for standard treatment for IV alteplase according to national guidelines27;
* Age of 18 years or older;
* Written informed consent (deferred).

Exclusion Criteria:

* Candidate for endovascular thrombectomy (i.e., a proximal intracranial large artery occlusion on CTA);
* Contra-indication for treatment with IV alteplase according to national guidelines27:

  * Arterial blood pressure exceeding 185/110 mmHg and not responding to treatment
  * Blood glucose less than 2.7 or over 22.2 mmol/L
  * Cerebral infarction in the previous 6 weeks with residual neurological deficit or signs of recent infarction on neuro-imaging
  * Head trauma in the previous 4 weeks
  * Major surgery or serious trauma in the previous 2 weeks
  * Gastrointestinal or urinary tract hemorrhage in the previous 2 weeks
  * Previous intracerebral hemorrhage
  * Use of anticoagulant with INR exceeding 1.7 or APTT exceeding 50 seconds
  * Known thrombocyte count less than 90 x 109 /L
  * Treatment with direct thrombin or factor X inhibitors, unless specific antidotum has been given, i.e. idarucizumab in case of dabigatran use.
* Pre-stroke disability which interferes with the assessment of functional outcome at 90 days, i.e. mRS > 2;
* Known pregnancy or if pregnancy cannot be excluded, i.e. did not have intercourse for > 6 months and no clinical signs of pregnancy, adequate use of any contraceptive method (e.g. intrauterine devices) or sterilization of the subject herself.
* Contra-indication for an MRI scan, i.e.:

  * an MRI incompatible pacemaker, ICD, pacing wires and loop records
  * metallic foreign bodies (e.g. intra-ocular)
  * prosthetic heart valves
  * blood vessel clips, coils or stents
  * an implanted electronic and/or magnetic implant or pump (e.g. neurostimulator)
  * cochlear implants
  * mechanical implants (implanted less than 6 weeks ago)
  * a copper intrauterine device
* Current Participation in any medical or surgical therapeutic trial other than DUMAS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2022-03-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Any intracranial hemorrhage according to the Heidelberg Bleeding Classification on MRI | 24-48 hours post-treatment

SECONDARY OUTCOMES:
Score on the National Institutes of Health Stroke Scale (NIHSS) | at 24 hours and 5-7 days post-treatment
  The NIHSS measures neurological deficit, ranging from 0 to 42, with higher scores indicating more severe neurological deficit.
Score on the modified Rankin Scale (mRS) | at 30 days
  The mRS is an ordinal scale ranging from 0 (no symptoms) to 6 (death) measuring the degree of disability or dependence in everyday life.
Infarct volume on MRI | at 24-48 hours
Change (pre-treatment vs. post-treatment) in abnormal perfusion volume based on TTP/MTT maps measured with CT perfusion at baseline and MRI | at 24-48 hours post treatment.
Secondary blood biomarkers of thrombolysis: d-dimer levels and fibrinogen levels. | 1 hour post-treatment, after 3 hours, and after 24 hours post-treatment,
Symptomatic intracranial hemorrhage (sICH) according to the Heidelberg Bleeding Classification | within 30 days
  sICH is defined as any intracranial hemorrhage followed by a neurological deterioration that can be attributed to that hemorrhage, defined as an increase of >= 4 points on the NIHSS or >= 2 points on a specific NIHSS item.
Death from any cause | Within 30 days
Major extracranial hemorrhage according to the ISTH criteria | within 24 hours of study drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- DUMAS trial office, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Ende NAM, Roozenbeek B, Smagge LEM, Luijten SPR, Aerden LAM, Kraayeveld P, van den Wijngaard IR, Lycklama A Nijeholt GJ, den Hertog HM, Flach HZ, Postma AA, Roosendaal SD, Krietemeijer GM, Yo LSF, de Maat MPM, Nieboer D, Del Zoppo GJ, Meurer WJ, Lingsma HF, van der Lugt A, Dippel DWJ; DUMAS Investigators. Safety and Efficacy of Dual Thrombolytic Therapy With Mutant Prourokinase and Small Bolus Alteplase for Ischemic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2023 Jul 1;80(7):714-722. doi: 10.1001/jamaneurol.2023.1262. PMID 37213122
- [Derived] van der Ende NAM, Roozenbeek B, Smagge LEM, Luijten SPR, Aerden LAM, Kraayeveld P, van den Wijngaard IR, Lycklama A Nijeholt GJ, den Hertog HM, Flach HZ, Wallace AC, Gurewich V, Del Zoppo GJ, Meurer WJ, Lingsma HF, van der Lugt A, Dippel DWJ; DUMAS Investigators. Dual thrombolytic therapy with mutant pro-urokinase and small bolus alteplase for ischemic stroke (DUMAS): study protocol for a multicenter randomized controlled phase II trial. Trials. 2022 Aug 9;23(1):641. doi: 10.1186/s13063-022-06596-z. PMID 35945566